CLINICAL TRIAL: NCT05042206
Title: An Open Label, Single-center, Phase 1 Study to Evaluate the Safety of Allogeneic Bone Marrow Derived Mesenchymal Stem Cell in Patients With Chronic Kidney Disease
Brief Title: Clinical Trial to Evaluate Safety of Allogeneic Bone Marrow Derived Mesenchymal Stem Cell in Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMC-P-12
Record Dates: First submitted 2021-08-25; First posted 2021-09-13 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease Stage 3B; Chronic Kidney Disease stage4
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cellgram-CKD (Experimental): Subjects receive a safety evaluation at 1 month, 3 months, 6 months, 9 months and 12 months after intravenous infusion of Cellgram-CKD 10mL at intervals of 2 weeks (14 days) 3 times.
  In the case of Cellgram-CKD, a milky white cell suspension solution is filled in a colorless and transparent plastic syringe, and the syringe tip is fixed with an obturator.
  Interventions: Biological: Cellgram-CKD

INTERVENTIONS:
Biological: Cellgram-CKD — Allogeneic bone marrow-derived mesenchymal stem cell therapy for the treatment of chronic kidney disease

SUMMARY:
This clinical trial is an open, single-center, phase 1 clinical trial to evaluate the safety of allogeneic bone marrow-derived mesenchymal stem cell injection in patients with chronic kidney disease.

The purpose is to evaluate the safety for 12 months after administration of Cellgram-CKD 3 times in 10 patients with chronic kidney disease.

DETAILED DESCRIPTION:
The screening test is performed after the clinical trial subject consents in writing to participate in the clinical trial.

Subjects who meet the inclusion/exclusion criteria are registered in the clinical trial, and Cellgram-CKD is injected intravenously by puncturing a vein with a needle. After injecting Cellgram-CKD three times at an interval of 2 weeks (14 days), the subject visits the testing institution at 1 month, 3 months, 6 months, 9 months and 12 months for safety evaluation.

However, since the safety of Cellgram-CKD has not been established, proceed as follows.

In the first 3 subjects who received the investigational product, if no adverse events of Grade 3 or higher according to the NCI-CTCAE related to the investigational product occur 14 days after the 1st and 2nd administration, and 1 month after the 3rd administration, the remaining subjects were sequentially treated. Register as a member and conduct clinical trials.

If an adverse event of Grade 3 or higher according to the NCI-CTCAE standard related to the test drug occurs in two of the first three subjects, the clinical trial is terminated early. is conducted by registering three additional test subjects in the same way as the first.

If one or more of the three subjects develops a Grade 3 or higher adverse event related to the investigational product, the clinical trial is terminated early, and the remaining subjects are treated only if all three subjects do not have a Grade 3 or higher adverse reaction related to the investigational product. Register to continue the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 19 and 79
* Those diagnosed with CKD stage 3b or 4 [eGFR 15 - 44 ml/min/1.73 m2] within 1 year before screening
* Those who voluntarily participated in the clinical trial and signed the Informed consent form

Exclusion Criteria:

* Those with severe cardiovascular disease (angina, myocardial infarction, unstable arrhythmia, heart failure, etc.) at the screening visit
* Those with the following medical history/comorbidities A. Gentamicin hypersensitivity reaction B. Solid cancer or malignant blood disease within 5 years prior to screening C. Clinically significant cognitive disorder, dementia or psychiatric disorder D. Alcohol or drug abuse E. Severe respiratory disease (COPD, asthma, pneumonia, pulmonary embolism, pneumothorax, etc.) F. Stroke G. Systemic autoimmune disease
* Those whose test results fall under the following at the screening visit A. Pathogenic microorganism test (Hbs Ag, HCV Ab, HIV Ab, Syphilis) positive B. Uncontrolled hypertension (systolic blood pressure >190 mmHg or diastolic blood pressure >100 mmHg) or hypotension (systolic blood pressure <90 mmHg or diastolic blood pressure <50 mmHg) C. AST and ALT ≥ upper limit of normal x 3.0 D. Total bilirubin ≥ upper limit of normal x 1.5
* At screening, those who have the following treatment history A. Those who are being treated for severe systemic infection B. Those who have been treated with immunosuppressant within 28 days prior to screening
* Those with a history of renal transplantation
* Those who have received dialysis within 3 months prior to the screening visit or who are planning to undergo dialysis during the clinical trial period
* Pregnant, lactating, or planning during clinical trials
* Those who do not agree to comply with the contraceptive method specified in this protocol during the clinical trial period
* Those who are receiving drugs that are expected to affect the results of this clinical trial when judged by the investigator
* Those who participated in other interventional clinical trials within 4 weeks prior to the screening visit and received investigational products/medical devices for investigational use or received procedures
* Those who have or are planning to administer other cell therapy products
* Those who are judged by the investigator to be inappropriate to participate in this clinical trial

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse event, and the level of the adverse event (AE) analyzed according to the Common Terminology Criteria for Adverse Event (CTCAE) (version 5.0) | Adverse events are collected from the first administration of the investigational product to 12 months after the third administration of the investigational product.
  The primary endpoint is an adverse event, and the level of the adverse event (AE) is analyzed according to the Common Terminology Criteria for Adverse Event (CTCAE) (version 5.0).

SECONDARY OUTCOMES:
Changes in eGFR | 1, 3, 6, 9, and 12 months of administration of the investigational product
  Changes in eGFR after 1, 3, 6, 9, and 12 months of administration of the investigational product compared to the baseline
Changes in BUN | 1, 3, 6, 9, and 12 months of administration of the investigational product
  Changes in BUN after 1, 3, 6, 9, and 12 months of administration of the investigational product compared to the baseline
Changes in Creatinine | 1, 3, 6, 9, and 12 months of administration of the investigational product
  Changes in Creatinine after 1, 3, 6, 9, and 12 months of administration of the investigational product compared to the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kim Hyosang, Principal Investigator — Asan Medical Center Nephrology
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No